CLINICAL TRIAL: NCT06011200
Title: A Randomized, Blinded, Comparable Vaccine-controlled Phase IIIb Clinical Trial to Evaluate the Safety and Immunogenicity of Meningococcal Polysaccharide Conjugate Vaccine, Group ACYW135 (CRM197 Vector), in a 4 to 6 Year-old Population
Brief Title: A Clinical Trial of ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector) in a 4 to 6 Year-old Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-MCVF-002
Record Dates: First submitted 2023-08-15; First posted 2023-08-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Epidemic Meningitis
Keywords: ACYW135; CRM197; Immunogenicity; Safety; 4~6 yearsof age
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197) (MCV4) (Experimental): Intramuscular injection, 0.5ml
  Interventions: Biological: MCV4
- ACYW135 Group Meningococcal Polysaccharide Vaccine (MSPV4) (Active Comparator): Subcutaneous injection, 0.5ml
  Interventions: Biological: MSPV4

INTERVENTIONS:
Biological: MCV4 — 1 dose of MCV4 on Day 0
  Arms: ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197) (MCV4)
Biological: MSPV4 — 1 dose of MSPV4 on Day 0
  Arms: ACYW135 Group Meningococcal Polysaccharide Vaccine (MSPV4)

SUMMARY:
The scientific name of meningococcus is Neisseria meningitidis (Nm), the causative agent of epidemic meningococcal meningitis (rheumatoid encephalitis), which colonizes the mucous membranes of the human nasopharynx or causes local infection and can cross the mucosal barrier to cause invasive bacteremia or epidemic meningococcal meningitis, meningococcus can often cause serious disease epidemics worldwide, the main clinical features of its infection are fever, rash and meningitis, the most common clinical manifestation is acute bacterial meningitis.

DETAILED DESCRIPTION:
The preventive measures for influenza are based on strengthening personal protection, vaccination, strengthening surveillance, early detection of patients, and active isolation and treatment. The immune response to meningococcal polysaccharide vaccine is weak in infants under 2 years of age, and only a transient immune response is produced. Numerous experiments have shown that the immunogenicity of polysaccharides is enhanced by binding to protein carriers, and a significant booster effect is produced. Meningococcal polysaccharide conjugate vaccine induces a good immune response in infants and children under 2 years of age and produces immune memory, which enhances the immune effect of the vaccine and can eliminate the carrier state of infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4~6 years old
* Complete at least two doses of basic immunization with polysaccharide influenza vaccine according to the immunization program
* The legal guardian or delegate has given informed consent, voluntarily signed the informed consent form, and is able to comply with the requirements of the clinical study protocol

Exclusion Criteria:

* Fever before inoculation, axillary temperature >37.0℃
* Previous history of immunization with meningococcal polysaccharide conjugate vaccine
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* History of epilepsy, convulsions or seizures or a history of psychiatric illness or family history
* Volunteers with current meningitis or a history of meningitis
* Volunteers treated with immunosuppressive therapy, cytotoxic therapy, glucocorticoids (excluding topical treatment, surface treatment for acute uncomplicated dermatitis, spray treatment for allergic rhinitis) within the past 6 months (<6 months)
* Received blood/plasma products or immunoglobulins within 60 days (<60 days) prior to study vaccination or planned to receive blood/plasma products or immunoglobulins throughout the study period
* Suffering from serious chronic diseases or conditions that are in a progressive stage and cannot be controlled smoothly, such as thyroid disease
* Volunteers with known or suspected diseases that are judged by the investigator to affect vaccination such as severe respiratory disease, acute infection or active chronic disease, severe cardiovascular disease, severe liver or kidney disease, malignancy, severe infectious or allergic skin disease
* History of serious adverse reactions associated with the vaccine and/or history of severe allergic reactions (e.g., systemic allergic reactions) to any component of the investigational vaccine
* Immunocompromised individuals with known or suspected immunodeficiency as determined by medical history and/or physical examination (e.g., malignancy, HIV, etc.)
* Bleeding constitution or condition associated with prolonged bleeding, investigators consider intramuscular injection to be contraindicated
* Live attenuated vaccine given within 14 days, other vaccines given within 7 days
* Participation in other studies involving interventions within 28 days (<28 days) prior to study entry and/or during study participation
* Other conditions judged by the investigator to be inappropriate for participation in this clinical trial

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of meningococcal antibodies to groups A, C, Y and W135 in all subjects 30 days after immunization | 30 days after immunization
Positive conversion rates of meningococcal antibodies to groups A, C, Y and W135 in all subjects 30 days after immunization | 30 days after immunization
Incidence of adverse reactions within 30 minutes after immunization in all subjects | Within 30 minutes after immunization
Incidence of adverse reactions/events within 7 days of immunization for all subjects | Within 7 days after immunization
Incidence of adverse reactions/events within 30 days of exemption for all subjects | Within 30 days of exemption

SECONDARY OUTCOMES:
Meningococcal positivity for groups A, C, Y, and W135 for all subjects 30 days after immunization | 30 days after immunization
Geometric mean growth multiplier (GMI) for all subjects 30 days after immunization | 30 days after immunization
Antibody titers ≥1:128 ratio for all subjects 30 days after immunization | 30 days after immunization
Meningococcal antibody positivity for groups A, C, Y and W135 at 90 and 180 days of exemption in 500 subjects | 90 and 180 days of exemption
GMT for groups A, C, Y and W135 at 90 and 180 days of exemption in 500 subjects | 90 and 180 days of exemption
GMI for groups A, C, Y and W135 at 90 and 180 days of exemption in 500 subjects | 90 and 180 days of exemption
Antibody titers ≥1:128 ratio for groups A, C, Y and W135 at 90 and 180 days of exemption in 500 subjects | 90 and 180 days of exemption
Incidence of serious adverse events (SAEs) within 180 days of exemption in all subjects | Within 180 days of exemption
All subjects were stratified into susceptible (<1:8) and non-susceptible (≥1:8) populations according to the 1:8 pre-immune antibody titer threshold | 30 days after immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Shanyang County Center for Disease Prevention and Control, Shanyang, Shaanxi, China